CLINICAL TRIAL: NCT06643832
Title: Spinal and Supra-spinal Modulation of Propofol Injection Pain by Rubbing and Distraction: A Randomized Controlled Study
Brief Title: Modulation of Propofol Injection Pain by Rubbing and Distraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, Lecturer of anesthesiology, surgical Intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR878/9/24
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-09

CONDITIONS: Propofol Injection; Pain; Rubbing; Distraction
Keywords: Pain, Modulation
MeSH Terms: conditions — Pain | interventions — Lidocaine; Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: open label for rubbing distraction group which is the novel approach to be tested in this trial (obviously, participant and pain assessor in the rubbing distraction group can not be blinded). however, lidocaine group and control group patients and their pain assessors are blinded to group assignment. so a final description of (partially blinded study) can be adopted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rubbing Distraction group (Experimental): rubbing and gently touching on proximal part of the intravenous injection site with the palm of the hand extending to the elbow. This will be started 5 seconds before propofol injection (not mixed with any drug) and continued until loss of consciousness. Also, a mobile video with duration of 10 seconds will be used for distraction and will be started 5 seconds before propofol injection so as to be ended at the time of first pain assessment.
  Interventions: Other: Rubbing Distraction
- Lidocaine group (Active Comparator): patients will receive intravenous propofol mixed with 2ml of lidocaine 2% (40mg) before injection.
  Interventions: Drug: Lidocaine (drug)
- Saline group (Placebo Comparator): patients will receive intravenous propofol not mixed with any drug (except for 2 ml of saline to ensure blindness of the outcome assessor).
  Interventions: Other: Saline

INTERVENTIONS:
Other: Rubbing Distraction — gently touching on proximal part of the IV injection site with the palm of the hand extending to the elbow. This will be started 5 seconds before propofol injection (not mixed with any drug) and continued until loss of consciousness. Also, a mobile video with duration of 10 seconds will be used for distraction and will be started 5 seconds before propofol injection so as to be ended at the time of first pain assessment.
  Arms: Rubbing Distraction group
Drug: Lidocaine (drug) — lidocaine will be used by mixing it with the propofol before intravenous injection
  Arms: Lidocaine group
Other: Saline — intravenous propofol will be given without mixing with any drug (except for 2 ml saline to ensure blindness of the outcome assessor).
  Arms: Saline group

SUMMARY:
This prospective randomized controlled study will be conducted to evaluate the effects of rubbing and distraction on the incidence and severity of propofol injection pain and compare them with the standard intravenous lidocaine method.

DETAILED DESCRIPTION:
Propofol has become one of the most common anesthetic agents used for sedation, induction, and maintenance of anesthesia because of its unique pharmacological properties. Pain during bolus injection is a major drawback with an incidence as high as 80%-90% in an untreated patient.

One of the most effective factors that alleviate the injection pain involves pretreatment with lidocaine.

Spinal modulation of pain is explained by the melzack gate control theory, it proposed that stimulation of A beta fibers by touch and vibration, modulate the dorsal horn "gate" and therefore the nociceptive input from the periphery could be reduced. (5) Regarding the use of this concept for managing propofol pain, only one study was conducted and revealed that rubbing didn't decrease the incidence but significantly decreased the severity of pain.

Distraction is a method of removing attention; so, it modifies cognitive pain perceptions by altering nociceptive responses and triggering an internal pain-suppressing system. Therefore, it causes a decrease in the activation of areas in the brain (e.g.: thalamus and insula) which contribute significantly to pain perception. we will combine rubbing and distraction, as methods for spinal and supra-spinal pain modulation, to evaluate their effects on propofol injection pain and compare them with the standard intravenous lidocaine method.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex
* American Society Anesthesiologists physical (ASA) status I-II
* age between 18-65 years old
* undergoing elective surgeries under general anesthesia using Propofol for anesthetic induction.

Exclusion Criteria:

* Allergy to experimental drugs
* Abuse of alcohol, analgesia, or sedative antidepressant
* Difficulty in communication
* Chronic pain syndromes, thrombophlebitis, neurological disease, and analgesic administration at the time of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of propofol injection pain | Pain will be evaluated every 5 seconds during the propofol injection until loss of concioussness. The highest pain score will be recorded
  Pain will be graded using a four-point scale: 0 = no pain, 1 = mild pain (pain reported only in response to questioning without any behavioral signs), 2 = moderate pain (pain reported in response to questioning and accompanied by a behavioral sign or pain reported spontaneously without questioning), and 3 = severe pain (i.e., strong vocal response or response accompanied by facial grimacing, arm withdrawal, or tears).

SECONDARY OUTCOMES:
Degree of pain | every 5 seconds during injection and the highest value will be recorded.
  Pain will be graded using a four-point scale: 0 = no pain, 1 = mild pain (pain reported only in response to questioning without any behavioral signs), 2 = moderate pain (pain reported in response to questioning and accompanied by a behavioral sign or pain reported spontaneously without questioning), and 3 = severe pain (i.e., strong vocal response or response accompanied by facial grimacing, arm withdrawal, or tears)
Recall of pain | 1 hour after surgery
  Patients who will report pain during propofol injection will be asked if they recalled this pain
adverse effects | 1 hour after surgery
  Like redness or edema will be examined at the site of propofol injection

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study
Access Criteria: The data will be available upon reasonable request from the corresponding author